CLINICAL TRIAL: NCT01904019
Title: Trapezio-metacarpal Arthroplasty: Comparison of ARPE Prosthesis With the Literature.
Brief Title: Comparison of ARPE Prosthesis With the Literature
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Collaborators: Biomet Belgium BVBA (Industry)
Responsible Party: Sponsor
Other Study IDs: ORTHO.CR.E16
Record Dates: First submitted 2013-06-19; First posted 2013-07-19 (Estimated); Results first posted 2021-08-23 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-09

CONDITIONS: Arthritis
Keywords: arthroplasty; trapezio-metacarpial
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is designed to document the objective and subjective measurements after trapeziometacarpal athroplasty with ARPE prosthesis and to compare those to literature values of outcome after trapeziectomy and trapeziectomy with ligament reconstruction and tendon interposition (LRTI), as published in a recent meta-analysis.

DETAILED DESCRIPTION:
The primary objective is to compare functional outcome at 3 years after trapezio-metarcarpal arthroplasty with trapeziectomy and trapeziectomy with ligament reconstruction and tendon interposition. Literature values obtained by a recently published meta analysis will be used.

The secondary objectives are:

* to compare functional outcome at 1 and at 5 years after trapezio-metarcarpal arthroplasty with trapeziectomy and trapeziectomy with ligament reconstruction and tendon interposition
* to determine pre- and post-operative HR QOL
* Incidence of radiolucencies at each follow up time point. Literature values from the same meta analysis will be used,

Patients will be assessed at preoperatively, and at 1, 3 and 5 years postoperatively. Measured Outcomes: grip strength, tip pinch strength, key pinch strength, pain, occurrence of adverse events, hand function.

ELIGIBILITY:
Inclusion/exclusion criteria are identical to those indications and contraindications stated in the package insert of the implant.

Inclusion Criteria:

* patients with trapezio-metacarpal arthritis Eaton Stage of trapezio-metacarpal arthritis: Stage II - IV
* patients willing to return for follow up evaluation.

Exclusion Criteria:

* local or systemic infections
* severe muscular, neurological or vascular deficiencies of the extremity involved
* bone destruction or poor bone to affect implant stability
* allergy to any of the components of the implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring a trapeziometacarpal arthroplasty to replace the trapeziometacarpal joint and restore its function.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-04; Primary Completion 2020-10 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederik VERSTREKEN, PhD, Principal Investigator — SPM Deurne
Locations (1):
- SPM Deurne, Deurne, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: According to the protocol, 100 subjects were to be enrolled. Due to the inclusion of 5 bilateral patients the actual number of participants is 95, but 100 implants were included in the study.
Units Other Than Participants: implants
Groups:
- ARPE Prosthesis: Single study patient cohort, including 95 patients (100 implants) receiving the cementless ARPE trapeziometacarpal prosthesis.
Period: Pre-operative
Arm/Group | ARPE Prosthesis
Started | 95; 100 implants
Completed | 95; 100 implants
Not Completed | 0; 0 implants
Period: 1 Year Follow-up
Arm/Group | ARPE Prosthesis
Started | 95; 100 implants
Completed | 86; 91 implants
Not Completed | 9; 9 implants
Not completed — Withdrawal by Subject | 4
Not completed — Impossibility to contact patient | 5
Period: 3 Year Follow-up
Arm/Group | ARPE Prosthesis
Started | 86; 91 implants
Completed | 71; 76 implants
Not Completed | 15; 15 implants
Not completed — Withdrawal by Subject | 1
Not completed — Impossibility to contact patient | 14
Period: 5 Year Follow-up
Arm/Group | ARPE Prosthesis
Started | 71; 76 implants
Completed | 65; 69 implants
Not Completed | 6; 7 implants
Not completed — Withdrawal by Subject | 2
Not completed — Impossibility to contact patient | 4

BASELINE CHARACTERISTICS:
Population: Number of Unilateral Patients: 90; Number of Bilateral Patients: 5.
Units Other Than Participants: implants
Arm/Group | ARPE Prosthesis
Number analyzed (Participants) | 95
Number analyzed (implants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (7.2)
Sex: Female, Male [Count of Units; unit: implants]
  Female | 87
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Surgery Side Distribution [Count of Units; unit: implants]
  Left | 59
  Right | 41
Weight Distribution [Mean (Standard Deviation); unit: kg] | 70.4 (14.5)
Height Distribution [Mean (Standard Deviation); unit: cm] | 165.3 (7.4)
Other Joint Involvement of the Hand [Count of Units; unit: implants]
  No | 31
  Yes | 69
Previous Hand Surgeries/Treatments on Affected Hand [Count of Units; unit: implants]
  No | 77
  Yes | 23
Trapezio Metacarpal Arthritis Disease Stage [Count of Units; unit: implants] — The Eaton radiographic classification system categorizes trapezio-metacarpal arthritis in 4 stages, with stage I being the better outcome and stage IV being the worst outcome. Stage I: slight joint space widening, normal articular contours; Stage II: Slight narrowing of joint space with osteophytes; Stage III: Marked narrowing of joint space with osteophytes, cystic changes, sclerotic bone; Stage IV: Complete deterioration of the joint, scaphotrapezial joint narrowed with sclerotic and cystic changes apparent.
  Only patients with Eaton Stages II to IV were included in this study.
  implants
    Stage II | 26
    Stage III | 68
    Stage IV | 6

OUTCOME MEASURES:

1. Primary Outcome: Grip Strength
Description: Grip strength is an indicator of muscle health in the hands and forearms and is measured with a hand-held dynamometer. The patients squeeze the dynamometer with all of their strength and the force applied is measured.
Time Frame: Pre-operative, 1, 3 and 5 years follow-up
Population: Due to the inclusion of 5 bilateral patients the actual number of participants is 95, but 100 implants were included in the study. The results are indicated per implant number.
Measure: Mean (Standard Deviation); unit: kg
Units Other Than Participants: implants
Arm/Group | ARPE Prosthesis
Number analyzed (Participants) | 95
Number analyzed (implants) | 100
kg
  Pre-operative | 17.8 (8.7)
  1 year follow-up: number analyzed (Participants) | 86
  1 year follow-up: number analyzed (implants) | 89
  1 year follow-up | 23.4 (9.2)
  3 years follow-up: number analyzed (Participants) | 71
  3 years follow-up: number analyzed (implants) | 75
  3 years follow-up | 24.7 (10.3)
  5 years follow-up: number analyzed (Participants) | 65
  5 years follow-up: number analyzed (implants) | 62
  5 years follow-up | 25 (8.9)

2. Primary Outcome: Key Pinch Strength
Description: Key pinch strength is an indicator of muscle health and measures the precision grip by using a pinch dynamometer. The device is placed between the radial side of the index finger and thumb and the force applied while the patients pinch as hard as possible is measured.
Time Frame: Pre-operative, 1, 3 and 5 years follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Units Other Than Participants: implants
Arm/Group | ARPE Prosthesis
Number analyzed (Participants) | 95
Number analyzed (implants) | 100
kg
  Pre-operative | 3.6 (2.1)
  1 year follow-up: number analyzed (Participants) | 86
  1 year follow-up: number analyzed (implants) | 87
  1 year follow-up | 5.8 (2.3)
  3 years follow-up: number analyzed (Participants) | 71
  3 years follow-up: number analyzed (implants) | 65
  3 years follow-up | 5.5 (2.1)
  5 years follow-up: number analyzed (Participants) | 65
  5 years follow-up: number analyzed (implants) | 62
  5 years follow-up | 5.9 (2.0)

3. Primary Outcome: Tip Pinch Strength
Description: Tip pinch strength is an indicator of muscle health and measures the precision grip by using a pinch dynamometer. The device is placed between the tip of the index finger and thumb and the force applied while the patients pinch as hard as possible is measured.
Time Frame: Pre-operative, 1, 3 and 5 years follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Units Other Than Participants: implants
Arm/Group | ARPE Prosthesis
Number analyzed (Participants) | 95
Number analyzed (implants) | 100
kg
  Pre-operative: number analyzed (implants) | 99
  Pre-operative | 2.7 (1.6)
  1 year follow-up: number analyzed (Participants) | 86
  1 year follow-up: number analyzed (implants) | 87
  1 year follow-up | 4.5 (1.8)
  3 years follow-up: number analyzed (Participants) | 71
  3 years follow-up: number analyzed (implants) | 66
  3 years follow-up | 4.6 (2)
  5 years follow-up: number analyzed (Participants) | 65
  5 years follow-up: number analyzed (implants) | 62
  5 years follow-up | 4.5 (1.5)

4. Primary Outcome: VAS Pain
Description: Pain level is collected with VAS (Visual Analog Scale): the patients are asked to mark their current pain level on a horizontal line containing values ranging from 0 (no pain) to 100 (very severe pain).
Time Frame: Pre-operative, 1, 3 and 5 years follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: implants
Arm/Group | ARPE Prosthesis
Number analyzed (Participants) | 95
Number analyzed (implants) | 100
score on a scale
  Pre-operative | 59.3 (19.5)
  1 year follow-up: number analyzed (Participants) | 86
  1 year follow-up: number analyzed (implants) | 91
  1 year follow-up | 11.1 (14.8)
  3 years follow-up: number analyzed (Participants) | 71
  3 years follow-up: number analyzed (implants) | 76
  3 years follow-up | 10.3 (19.6)
  5 years follow-up: number analyzed (Participants) | 65
  5 years follow-up: number analyzed (implants) | 69
  5 years follow-up | 7.1 (15.1)

5. Secondary Outcome: Motion - ROM Measurement - Radial Abduction
Description: The range of motion (ROM) is the extent of movement of a joint and indicates the range through which the joint can be moved. ROM in radial abduction is measured while the patients move the thumb in parallel to the palm.
Time Frame: Pre-operative, 1, 3 and 5 years follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: implants
Arm/Group | ARPE Prosthesis
Number analyzed (Participants) | 95
Number analyzed (implants) | 100
degrees
  Pre-operative | 41.5 (7.1)
  1 year follow-up: number analyzed (Participants) | 86
  1 year follow-up: number analyzed (implants) | 90
  1 year follow-up | 53.1 (37.8)
  3 years follow-up: number analyzed (Participants) | 71
  3 years follow-up: number analyzed (implants) | 76
  3 years follow-up | 47.5 (6.1)
  5 years follow-up: number analyzed (Participants) | 65
  5 years follow-up: number analyzed (implants) | 62
  5 years follow-up | 43.8 (9.9)

6. Secondary Outcome: Motion - ROM Measurement - Palmar Abduction
Description: The range of motion (ROM) is the extent of movement of a joint and indicates the range through which the joint can be moved. The ROM in palmar abduction is measured while the patients move the thumb perpendicularly to the palm.
Time Frame: Pre-operative, 1, 3 and 5 years follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: implants
Arm/Group | ARPE Prosthesis
Number analyzed (Participants) | 95
Number analyzed (implants) | 100
degrees
  Pre-operative | 43.2 (5.8)
  1 year follow-up: number analyzed (Participants) | 86
  1 year follow-up: number analyzed (implants) | 90
  1 year follow-up | 48.1 (6.4)
  3 years follow-up: number analyzed (Participants) | 71
  3 years follow-up: number analyzed (implants) | 76
  3 years follow-up | 47.8 (5.9)
  5 years follow-up: number analyzed (Participants) | 65
  5 years follow-up: number analyzed (implants) | 62
  5 years follow-up | 43.4 (8.4)

7. Secondary Outcome: EQ-5D - Health Status Score
Description: EQ-5D is a standardized instrument for measuring the health-related quality of life, which assesses health status in terms of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each question has five levels of response (no problems, slight problems, moderate problems, severe problems, extreme problems/unable to), which are singularly rated and then combined into a health status score. The health status score ranges from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility.
Time Frame: Pre-operative, 1, 3 and 5 years follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: implants
Arm/Group | ARPE Prosthesis
Number analyzed (Participants) | 95
Number analyzed (implants) | 100
score on a scale
  Pre-operative | 0.4 (0.3)
  1 year follow-up: number analyzed (Participants) | 86
  1 year follow-up: number analyzed (implants) | 91
  1 year follow-up | 0.8 (0.3)
  3 year follow-up: number analyzed (Participants) | 71
  3 year follow-up: number analyzed (implants) | 76
  3 year follow-up | 0.8 (0.3)
  5 year follow-up: number analyzed (Participants) | 65
  5 year follow-up: number analyzed (implants) | 69
  5 year follow-up | 0.8 (0.3)

8. Secondary Outcome: EQ-5D - VAS Score
Description: The second part of the EQ-5D questionnaire consists of a visual analogue scale (VAS) on which the patient rates his/her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).
Time Frame: Pre-operative, 1, 3 and 5 years follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: implants
Arm/Group | ARPE Prosthesis
Number analyzed (Participants) | 95
Number analyzed (implants) | 100
score on a scale
  Pre-operative | 72.7 (15.8)
  1 year follow-up: number analyzed (Participants) | 86
  1 year follow-up: number analyzed (implants) | 91
  1 year follow-up | 74.1 (19.5)
  3 years follow-up: number analyzed (Participants) | 71
  3 years follow-up: number analyzed (implants) | 76
  3 years follow-up | 77.9 (15.7)
  5 years follow-up: number analyzed (Participants) | 65
  5 years follow-up: number analyzed (implants) | 69
  5 years follow-up | 76.2 (17.2)

9. Secondary Outcome: Number of Implants With Visible Radiolucency Line Around the Implanted Prosthesis
Description: Radiolucency lines are radiolucent gaps visible in the radiographic images between the prosthesis and the bone, which presence is commonly associated with early failure of the implantation, eventually leading to the loosening of the prosthesis. Every radiography taken at each follow-up time point was assessed to evaluate whether there are visible radiolucency lines around the implanted prosthesis and the number of implants with visible radiolucency lines is here reported.
Time Frame: 1, 3 and 5 years follow-up
Population: Due to the inclusion of 5 bilateral patients the actual number of participants is 95, but 100 implants were included in the study. The results are indicated per implant number. There were no radiolucency lines reported for any of the patients included in the study at any time point.
Measure: Count of Units; unit: implants
Units Other Than Participants: implants
Arm/Group | ARPE Prosthesis
Number analyzed (Participants) | 95
Number analyzed (implants) | 100
implants
  1 years follow-up: number analyzed (Participants) | 86
  1 years follow-up: number analyzed (implants) | 91
  1 years follow-up | 0
  3 years follow-up: number analyzed (Participants) | 71
  3 years follow-up: number analyzed (implants) | 76
  3 years follow-up | 0
  5 years follow-up: number analyzed (Participants) | 65
  5 years follow-up: number analyzed (implants) | 69
  5 years follow-up | 0

10. Secondary Outcome: Hand Function: DASH Questionnaire - Disability
Description: The DASH (Disabilities of the Arm, Shoulder and Hand) Questionnaire outcome measure is a 30-item, self-report questionnaire designed to assess the patients' health status during the previous week by asking to rate their ability to perform various daily activities. The questions are grouped in 3 categories: disability, work and sport, of which work and sport are optional.
  The score ranges from 0 (no disability) to 100 (most severe disability), with higher scores indicating a greater level of disability and severity, whereas lower scores indicate a lower level of disability.
Time Frame: Pre-operative, 1, 3 and 5 years follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: implants
Arm/Group | ARPE Prosthesis
Number analyzed (Participants) | 95
Number analyzed (implants) | 100
score on a scale
  Pre-operative | 41.7 (17.9)
  1 year follow-up: number analyzed (Participants) | 86
  1 year follow-up: number analyzed (implants) | 91
  1 year follow-up | 10.6 (14.3)
  3 year follow-up: number analyzed (Participants) | 71
  3 year follow-up: number analyzed (implants) | 76
  3 year follow-up | 10.2 (14.2)
  5 year follow-up: number analyzed (Participants) | 65
  5 year follow-up: number analyzed (implants) | 69
  5 year follow-up | 8.5 (11.8)

11. Secondary Outcome: Hand Function: DASH Questionnaire - Work
Description: as for outcome 10
Time Frame: Pre-operative, 1, 3 and 5 years follow-up
Population: Due to the inclusion of 5 bilateral patients the actual number of participants is 95, but 100 implants were included in the study. The results are indicated per implant number. The Work category is optional.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: implants
Arm/Group | ARPE Prosthesis
Number analyzed (Participants) | 95
Number analyzed (implants) | 100
score on a scale
  Pre-operative: number analyzed (implants) | 63
  Pre-operative | 46.1 (25.9)
  1 year follow-up: number analyzed (Participants) | 86
  1 year follow-up: number analyzed (implants) | 59
  1 year follow-up | 11.1 (17.2)
  3 year follow-up: number analyzed (Participants) | 71
  3 year follow-up: number analyzed (implants) | 28
  3 year follow-up | 7.8 (16.5)
  5 year follow-up: number analyzed (Participants) | 65
  5 year follow-up: number analyzed (implants) | 15
  5 year follow-up | 5.8 (13.5)

12. Secondary Outcome: Hand Function: DASH Questionnaire - Sport
Description: as for outcome 10
Time Frame: Pre-operative, 1, 3 and 5 years follow-up
Population: Due to the inclusion of 5 bilateral patients the actual number of participants is 95, but 100 implants were included in the study. The results are indicated per implant number. The Sports category is optional.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: implants
Arm/Group | ARPE Prosthesis
Number analyzed (Participants) | 95
Number analyzed (implants) | 100
score on a scale
  Pre-operative: number analyzed (implants) | 33
  Pre-operative | 48.7 (32.4)
  1 year follow-up: number analyzed (Participants) | 86
  1 year follow-up: number analyzed (implants) | 27
  1 year follow-up | 6.7 (13.4)
  3 year follow-up: number analyzed (Participants) | 71
  3 year follow-up: number analyzed (implants) | 21
  3 year follow-up | 10.1 (21.8)
  5 year follow-up: number analyzed (Participants) | 65
  5 year follow-up: number analyzed (implants) | 14
  5 year follow-up | 2.2 (5.8)

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events from the date each subject was implanted up to 5 years after surgery, when the last follow-up was performed and patients completed the study.
Description: Adverse events were collected in an Adverse Event Form, which gathers information on the date of occurrence, the nature of the adverse event, whether the device was involved, which treatment was used and the treatment outcome.
Arm/Group | ARPE Prosthesis
All-Cause Mortality (participants affected / at risk) | 0/95
Serious Adverse Events (participants affected / at risk) | 17/95
Other Adverse Events (participants affected / at risk) | 19/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARPE Prosthesis (N=95)
Prosthesis luxation (Musculoskeletal and connective tissue disorders) | 5 (6) — Device-related SAE
Hip replacement (Surgical and medical procedures) | 2 (2) — Resolved with surgery
Anaphylactic shock (General disorders) | 1 (1) — To unknown medication, resolved with hospitalization
Discectomy (Surgical and medical procedures) | 1 (1)
Malnutrition (General disorders) | 1 (1) — Resolved with hospitalization and diet
Heart arrhythmia (Cardiac disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gonarthrosis (Surgical and medical procedures) | 1 (1) — Resolved with surgery
Neck problems (Musculoskeletal and connective tissue disorders) | 1 (1)
Prostate hypertrophy (Reproductive system and breast disorders) | 1 (1) — Resolved with surgery
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Resolved with surgery
Bladder prolapse (Renal and urinary disorders) | 1 (1) — Resolved with surgery
Gastric bleeding (Gastrointestinal disorders) | 1 (1)
Rizarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) — In contralateral thumb, resolved with surgery
Cuff tear shoulder (Surgical and medical procedures) | 1 (1) — Resolved with surgery
Fracture of pseudoarthrosis radius (Surgical and medical procedures) | 1 (1) — Resolved with surgery
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARPE Prosthesis (N=95)
Thumb pain (Musculoskeletal and connective tissue disorders) | 3 (3) — Device-related
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 11 (13) — De Quervain tenosynovitis
Thumb and/or wrist pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Caused by overload; device-related therefore reported even if <1% frequency
Carpal tunnel (Musculoskeletal and connective tissue disorders) | 4 (5)
Thumb infection (Infections and infestations) | 1 (2)
Arthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) — STT arthrosis and arthrosis in midcarpal and radiocarpal; device-related therefore reported even if <1% frequency

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-11-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT01904019/Prot_SAP_001.pdf